CLINICAL TRIAL: NCT01603225
Title: The Use of Transcranial Direct Current Stimulation (tDCS) to Improve Communicative Efforts, Speech, Language and Related Cognitive Functions in Individuals With Autism
Brief Title: Transcranial Direct Current Stimulation and Autism
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00042345
Record Dates: First submitted 2012-05-17; First posted 2012-05-22 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; tDCS
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Autism: Individuals with autism will have either Anodal, Cathodal, or Sham Transcranial Direct Current Stimulation (tDCS).
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Delivery of transcranial direct current stimulation for 30-60 minutes or sham stimulation.This will be administered by two or more similar devices.

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve certain mental abilities, such as speech, language and other efforts at communication in individuals with autism.

In this research, battery powered device is used to deliver very weak electrical current to the surface of the scalp while participants are involved in tasks aimed at training or measuring communicative efforts, speech, language or related cognitive functions. Our aim is to find out whether tDCS will improve these mental abilities.

DETAILED DESCRIPTION:
Participants in the study will be asked to do the following things:

* Grant permission for the researchers to view medical/psychological and/or educational and/or speech records associated with the diagnosis of low-functioning autism.
* Complete a questionnaire and provide a health history.
* Complete evaluations by our study team to assess the diagnosis and gain a clearer understanding of the participant's current functioning.
* Give permission to audio and video-tape test sessions for later scoring and observation.
* Give permission to audio or video-tape in the classroom or home environment using non-intrusive audio-visual recording devices.
* Complete several tasks and training interventions that involve such things as learning new words or pictures, saying words out loud, or naming objects.
* Participate in an eye tracking study while completing a task on the computer which involves wearing a headband, attached by a velcro fastener, which contains a magnetic sensor. This equipment allows us to track the position of the head in order to record more accurate measurements. It is used with eye tracking equipment which measures the gaze on a set point on a computer screen. The equipment poses no risk and is non-invasive.
* Participate in computerized tasks while monitoring brain responses that are a direct result of a thought or perception. In order to monitor these responses, electrodes would be placed over various points on your scalp. The electrodes will record the on-going activity of the brain; it does not produce or introduce any electrical activity. The equipment poses no risk and is non-invasive.
* Wear electrodes that will be placed on the scalp with a large rubberized band. These electrodes will administer very weak electrical current (tDCS) from a battery powered device for 20 to 60 minutes.

The experimental sessions will last about 1 hour and participants may be asked to have more than one testing session in a day or to return for additional sessions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism or related conditions
* Identified language deficit(s) and/or other cognitive or behavioral impairments (which will be specific to each sub-study)
* Adequate ability to perform the research tasks set for the individual's particular level of performance

Exclusion Criteria:

* Peripheral blindness or deafness
* Any implanted metal device (precludes use of tDCS)
* Any implanted cardiac pacemaker

Ages: 14 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The experimental group will consist of adults with autism (n=40). Participants will be 18-79 years of age, diagnosed with autism by independent clinicians and confirmed by formal assessment (e.g., CDI, ADOS, Bayley, Sensory Profile), and with receptive and expressive vocabulary levels of ≥ 3 years age-equivalent, as assessed by standardized measures. Additionally, the Autism Diagnostic Interview will be administered to caregivers in order to appropriately identify specific areas (regarding speech, language and cognition) in which participants are experiencing the most difficulty.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-26 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Picture naming accuracy | 10 minutes
  Oral naming of visually-presented pictures, measured in terms of accuracy. (Note: this task may not be included in the final design, nor given to all subjects)
Picture naming speed | 10 minutes
  Oral naming of visually-presented pictures, measured in terms of speed (milliseconds). (Note: this task may not be included in the final design, nor given to all subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Gordon, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Neurology; Cognitive Neurology/Neuropsychology, Baltimore, Maryland, United States